CLINICAL TRIAL: NCT00922857
Title: Influence of Muscular Atrophy on Biological and Functional Benefit of Respiratory Rehabilitation in Patients With Chronic Respiratory Failure
Acronym: INSPIRE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0408079; 2005/0023 (Other: DGS)
Record Dates: First submitted 2009-06-16; First posted 2009-06-17 (Estimated); Last update posted 2014-07-24 (Estimated); Status verified 2014-07

CONDITIONS: Respiratory Insufficiency
Keywords: Respiratory Insufficiency; Muscular Atrophy; Respiratory rehabilitation
MeSH Terms: conditions — Respiratory Insufficiency; Muscular Atrophy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Respiratory rehabilitation (Experimental)
  Interventions: Procedure: Respiratory rehabilitation

INTERVENTIONS:
Procedure: Respiratory rehabilitation — The training begins 5 days after the initial assessment. It consists of 3 weekly sessions for 8 consecutive weeks, including the following activities interspersed with periods of rest, according to the needs of patients

SUMMARY:
The prevalence of chronic respiratory failure (CRF) is increasing worldwide and will become the 3rd cause of death by 2020. At the stage of the disease requiring ventilatory assistance, this relates to 50,000 patients in France, life expectancy is very limited, and quality of life is poor.

CRF led to a reduction in muscle mass, which is found in 35 and 55% of patients, in some to a profound cachexia. A reduced fat free mass (FFM) is a factor associated with a poor tolerance to exercise and an halved survival. The exact causes and mechanisms leading to cachexia are not yet established. Recently, a chronic inflammatory condition has been quoted as a putative cause. This chronic inflammation would involve the molecular mechanisms leading to poor regulation of the balance of synthesis / protein degradation in muscle. A decrease in plasma and muscle amino acids was found among patients with a low FFM.. In addition, a decrease of plasma levels of some anabolic hormones, GH and androgens or IGF-1 has been found that could explain a lack of protein synthesis.

It is now well established that respiratory rehabilitation, including a program of exercise reconditioning, increases tolerance to exercise and improve the quality of life. Besides the classical type of endurance exercises stimulating the cardio-respiratory system, it is suggested to add resistance exercises. Several studies have reported the benefit of this strategy but the link with intracellular molecular pathways has not been described; moreover, it is unknown whether the existence of an initial muscular atrophy influences the gain in muscle strength/mass.

DETAILED DESCRIPTION:
We therefore propose to explore the effect of a rehabilitation program including endurance and resistance exercises on muscle biopsies.

The present study should help to know the molecular pathways implicated in muscle atrophy in CRF patients and to assess their evolution with rehabilitation. This could lead to individualized recommendation for exercise program according to the muscle mass of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Prescription of an exercise training program as part of a respiratory rehabilitation
* Existence of an obstructive ventilatory deficit
* Signature of written consent

Exclusion Criteria:

* Exacerbation of COPD
* Patient with a long-term oxygen therapy
* Active smoker
* Lower limb locomotor limitation preventing to achieve the full respiratory rehabilitation program
* Lower limbs arteritis
* Myocardial infarction or pulmonary embolism of less than 3 months
* Long term anticoagulant
* Type 1 diabetes

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2005-04; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Gain in exercise tolerance (relative variation of the 6 min walking distance and maximal exercise capacity on bicycle (peak VO2) combined with activation of the pathway for muscle protein synthesis | before and at the outcome of the reconditioning program in the effort

SECONDARY OUTCOMES:
Quality of life assessed by questionnaire | before and at the outcome of the reconditioning program in the effort

CONTACTS AND LOCATIONS:
Overall Officials: Frédéric COSTES, MD PhD, Principal Investigator — CHU de Saint-Etienne
Locations (1):
- CHU de Saint-Etienne, Saint-Etienne, France

REFERENCES:
- [Derived] Costes F, Gosker H, Feasson L, Desgeorges M, Kelders M, Castells J, Schols A, Freyssenet D. Impaired exercise training-induced muscle fiber hypertrophy and Akt/mTOR pathway activation in hypoxemic patients with COPD. J Appl Physiol (1985). 2015 Apr 15;118(8):1040-9. doi: 10.1152/japplphysiol.00557.2014. Epub 2015 Feb 19. PMID 25701004